CLINICAL TRIAL: NCT00958152
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Sequential-group, Multiple-dose, Drug-drug Interaction Study of VCH-222 and Telaprevir in Healthy Subjects
Brief Title: Drug-Drug Interaction Study of VCH-222 and Telaprevir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Robert Kauffman, M.D., Ph.D., Vertex Pharmaceuticals Incorporated
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: VX09-222-002
Record Dates: First submitted 2009-08-06; First posted 2009-08-13 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Hepatitis C
Keywords: VX-950; VX-222; STAT-C
MeSH Terms: conditions — Hepatitis C | interventions — lomibuvir; telaprevir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: VCH-222; Drug: telaprevir
- Cohort 2 (Experimental)
  Interventions: Drug: VCH-222; Drug: telaprevir
- Cohort 3 (Experimental)
  Interventions: Drug: VCH-222; Drug: telaprevir

INTERVENTIONS:
Drug: VCH-222 — Capsules, Oral, 400 mg, q12h, Days 1-10 and Days 28-37
  Arms: Cohort 1
Drug: VCH-222 — Capsules, Oral, 750 mg, q12h, Days 1-10 and Days 28-37
  Arms: Cohort 2
Drug: VCH-222 — Capsules, Oral, 1000 mg, q12h, Days 1-10 and Days 28-37
  Arms: Cohort 3
Drug: telaprevir — Tablet, Oral, 1125 mg, q12h, Days 18-37

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics, safety, and tolerability of the co-administration of VCH-222 and telaprevir in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, and/or healthy females of non-childbearing potential, aged 18 to 55 years (inclusive)
* Body mass index (BMI) between 18 and 31 kg/m2 (inclusive) and weight > 50 kg

Exclusion Criteria:

* Women of child bearing potential
* Subjects positive for Hepatitis B, Hepatitis C, or HIV
* Subjects who have participated in a clinical study involving administration of an investigational drug within 2 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability based on vital signs, 12-lead electrocardiograms (ECGs), physical examination, laboratory assessments, and adverse events | Day 47 safety assessment

SECONDARY OUTCOMES:
Pharmacokinetic parameters (Cmax, tmax, C12 h, Cmin, and AUC0-12 h) of VCH-222 at steady-state in plasma in the presence and absence of telaprevir at steady-state | Day 37 pharmacokinetic assessment
Pharmacokinetics parameters (Cmax, tmax, C12 h, Cmin, and AUC0-12 h) of telaprevir at steady-state in plasma in the presence and absence of VCH-222 at steady-state | Day 37 pharmacokinetic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (1):
- Christchurch, New Zealand